CLINICAL TRIAL: NCT06339528
Title: Potential of Vojta's Reflex Locomotion as a Pre/Induction Method for Uterine Activity: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jan Zapletal, Medical Doctor, Department of Obstetrics and Gynecology, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-VPl421012021
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Induced Vaginal Delivery
Keywords: Vojta's Reflex Locomotion; Induction of Labor; Delivery; Term pregnancy

STUDY DESIGN:
Intervention Model Description: A total of 40 pregnant patients between 40+0 to 41+0 weeks of gestational age were randomly selected for this study. Stimulation of trigger zones according to Vojta's therapy was applied to 20 of them by a team of licensed physiotherapists while a control group received a sham stimulation carried out by physicians. Cardiotocographic (CTG) recordings were conducted right before and immediately after stimulation. CTG recordings were subsequently blindly evaluated by 2 independent obstetricians.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Stimulation of trigger zones according to Vojta's therapy was applied to 20 of them by a team of licensed physiotherapists while a control group received a sham stimulation carried out by physicians. Cardiotocographic (CTG) recordings were conducted right before and immediately after stimulation. CTG recordings were subsequently blindly evaluated by 2 independent obstetricians. Patients did not know if clinician have skills to stimulate properly according to the Vojta's Reflex Locomotion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group stimulated according to the Vojta's Reflex Locomotion (Experimental): Stimulation of trigger zones according to Vojta was applied to 20 of them by a team of licensed physiotherapists.
  Interventions: Procedure: Vojta's Reflex Locomotion
- control group received a sham stimulation carried out by physicians (Placebo Comparator): Control group received a sham stimulation carried out by physicians.
  Interventions: Procedure: Sham stimulation

INTERVENTIONS:
Procedure: Vojta's Reflex Locomotion — Reflex locomotion according to Vojta's therapy is a neurorehabilitative concept originally used for diagnostics and treatment of infants who were at risk of non-physiological psychomotor development, especially spastic cerebral palsy. This concept utilizes stimulation of specific zones described by Vojta to evoke global motor and non-motor response.
  Trigger zones are specific body zones that are stimulated with pressure during reflex locomotion stimulation. They are pressure stimulated in order to induce reflex response. Variations of stimulation of different trigger zones (spatial summation) causes multiplication of afferent impulses. Sufficiently long stimulation of trigger zones (temporal summation) induces isometric contraction in muscle groups described by Vojta.
  Other Names: Vojta's method; Vojta's therapy
  Arms: group stimulated according to the Vojta's Reflex Locomotion
Procedure: Sham stimulation — Control group received sham stimulation by physicians at zones outside of the pressure zones, specifically 4-5 cm above the patella and on the lateral malleolus.
  Arms: control group received a sham stimulation carried out by physicians

SUMMARY:
The Vojta's method is neurophysiological rehabilitation method used to support and induce reflex responses of locomotor and vegetative system. It uses involuntary motor reaction of the body during pressure stimulation of so-called trigger zones. Pregnancy is currently considered a contraindication for using Vojta's therapy to potential risks of inducing regular uterine activity and risk of delivery. The aim of the study is to evaluate changes in uterine activity and also explore the possibility of using this method as a new approach for pre/induction of delivery.

DETAILED DESCRIPTION:
Reflex locomotion according to Vojta's therapy is a neurorehabilitative concept originally used for diagnostics and treatment of infants who were at risk of non-physiological psychomotor development, especially spastic cerebral palsy. This concept utilizes stimulation of specific zones described by Vojta to evoke global motor and non-motor response.

Trigger zones are specific body zones that are stimulated with pressure during reflex locomotion stimulation.

According to the author of Vojta's reflex locomotion (VRL) - Václav Vojta, there are 10 trigger zones on human body. These trigger zones are pressure stimulated in order to induce reflex response. On upper and lower extremities periosteum is stimulated by pressure stimulation of trigger zones. During pressure stimulation of trigger zones on trunk autochthone musculature is stimulated. By stimulation of trigger zones located on joints, ligaments and joint surfaces are stimulated. Vojta's method uses spatial and temporal summation of signals of stimulated trigger zones. Variations of stimulation of different trigger zones (spatial summation) causes multiplication of afferent impulses. Sufficiently long stimulation of trigger zones (temporal summation) induces isometric contraction in muscle groups described by Vojta.

Motor response to trigger zones stimulation is involuntary and it manifests as a symmetrical as well as asymmetrical movement of the limbs, trunk, neck and head. These movements are sorted into two main movement complexes - reflex creeping and reflex rolling.

There are several different indications that may be a reason for using VRL. Some of the main indications in children include: cerebral palsy, hypotonia, hypertonia, coordination disorders, scoliosis and spinal cord injury. In adults, VRL is used as a treatment in many diseases of musculoskeletal apparatus, e.g.: vertebrogenic disorders, condition after stroke, muscular disorders and others.

Several contraindications to the use of VRL should be considered when planning the treatment. Some of the main contraindications include: acute inflammation or infection, severe cardiovascular disease, acute joint or muscle pain or injury, severe neurological diseases, acute respiratory, and pregnancy for the risk of inducing uterine activity.

In obstetrics the two primary methods of inducing labor are pharmacological and non- pharmacological. The most commonly used non-pharmacological methods include cervical ripening using a balloon catheter with membrane sweeping efficient at 20% of patients or amniotomy, which can reduce duration of labor by approximately 2 hours.

This study aims to investigate the potential of VRL in initiating uterine activity and explore its feasibility as a new pre/induction method.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancy between 40+0 and 41+0 weeks of gestational age
* physiological evaluation of the pregnancy
* cervix score of at least 6
* signed written consent after a detailed explanation of the potentional benefits and risks associated with the simulation method.

Exclusion Criteria:

* pathological pregnancy
* cervix score less then 6

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Cardiotocographic (CTG) recordings - | right before and immediately after stimulation
  . Standard parameters such as basal rate, presence of accelerations and decelerations and variability of recording were evaluated in the cardiography recording. The tocographic record evaluated the presence of uterine activity, its intensity and regularity. CTG recordings were subsequently evaluated by 2 independent obstetricians.
subjective perception during stimulation | immediately after stimulation
  Non validated questionnaires were distributed to all the participants asking about subjective perception of contractions, body movement, breathing, pleasantness and pain. A scale from 1 to 10 for perception was made where 1 meant that stimulation was very pleasant and 10 was extremely unpleasant.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milan M, Jan Z, Vit D, Nikola J, Barbora S, Anna B, Radovan V, Lukas R, Michael HJ, Tereza N. Safety of Vojta's reflex locomotion in term pregnancy: a randomized controlled pilot study of uterine activity and labor onset. Sci Rep. 2026 Jan 15;16(1):2095. doi: 10.1038/s41598-025-31871-9. PMID 41540080